CLINICAL TRIAL: NCT03480126
Title: Assessing the Efficacy of Herbal Teas on Bone Health in an Osteopenic Population: OsTea
Brief Title: Herbal Teas on Bone Health in an Osteopenic Population
Acronym: OsTea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paula Witt-Enderby (Other)
Collaborators: Duquesne University (Other)
Responsible Party: Sponsor-Investigator, Paula Witt-Enderby, Professor of Pharmacology, Duquesne University
Organization: Duquesne University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018/02/7
Record Dates: First submitted 2018-02-28; First posted 2018-03-29 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Teas, Herbal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Herbal Tea 1 (Placebo Comparator): Placebo Tea should will be ingested 3 times per day for 3 months
  Interventions: Other: Herbal Teas
- Herbal Tea 2 (Experimental): Experimental Herbal Tea A will be ingested 3 times per day for 3 months
  Interventions: Other: Herbal Teas
- Herbal Tea 3 (Experimental): Experimental Herbal Tea B will be ingested 3 times per day for 3 months
  Interventions: Other: Herbal Teas
- Herbal Tea 4 (Experimental): Experimental Herbal Tea C will be ingested 3 times per day for 3 months
  Interventions: Other: Herbal Teas

INTERVENTIONS:
Other: Herbal Teas — Steeped tea ingested 3 times a day for 3 mos

SUMMARY:
The project goal is to identify if herbal teas consumed three times per day over a period of three months can improve these markers of bone health as well as improve quality of life (QOL) compared to women taking placebo by increasing osteoblast activity, decreasing osteoclast activity, increasing nocturnal melatonin levels and by decreasing C-reactive protein (CRP) and cortisol levels. Our central hypothesis is that these herbal teas will improve both objective and subjective measures of bone health in a population with osteopenia not taking this regimen by reducing osteoclast activity and increasing osteoblast activity and by reducing stress and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* male or female with osteopenia (T-score between -1.0 and -2.5)
* at least 18 years of age
* must be willing to drink tea three times a day for 3 months
* must also be willing to come to the study location on 4 occasions (baseline, end of month 1, end of month 2, and end of month 3),
* must also be willing to come to the study location to provide urinary, salivary and fecal samples on 2 occasions (baseline and at the end of month 3),
* must also be willing to come to the study location to have their blood pressure taken on 4 occasions (baseline, end of month 1, end of month 2, and end of month 3)
* must be willing to come to the study location to complete questionnaires on 2 occasions (baseline and at the end of month 3)
* must be willing to maintain daily diary for 4 months.

Exclusion Criteria:

* Women or men with osteoporosis
* Women or men with osteopenia due to hyperparathyroidism, multiple myeloma, metastatic bone disease, chronic steroid use
* Women or men who are on any bone therapies (i.e. bisphosphonates, selective estrogen receptor modulators, hormone therapy, teriparatide, and denosumab)
* Women or men with chronic obstructive pulmonary disease (COPD)
* Women or men who smoke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
The Effect of 3 month Herbal Tea on Changes in Human Type 1 Collagen C-telopeptide (CTx) levels | 3 months
  Urinary CTx levels will be measured at times month 0 (baseline) and month 3
The Effect of 3 month Herbal Tea on Changes in Human Procollagen Type 1 Intact N-terminal Propeptide (Total P1NP) levels | 3 months
  Urinary P1NP levels will be measured at times month 0 (baseline) and month 3
The Effect of 3 month Herbal Tea on Changes in the Ratio of CTx:P1NP | 3 months
  Urinary CTx:P1NP levels will be measured at times month 0 (baseline) and month 3

CONTACTS AND LOCATIONS:
Overall Officials: Paula A Witt-Enderby, PhD, Principal Investigator — Duquesne University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study assessing the efficacy of herbal teas on bone health and quality of life in a population with osteopenia: rooibos actions on melatonin and tulsi actions on quality of life. — https://www.melatonin-research.net/index.php/MR/article/view/135/778